CLINICAL TRIAL: NCT02708550
Title: Deltagerinvolverende Intervention for Bedre Brug af hjælpemidler i hospitalsvæsenet
Brief Title: Participatory Organizational Intervention for Improved Use of Assistive Devices for Patient Handling
Acronym: IRMA12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRMA12
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Disorders; Occupational Injuries
MeSH Terms: conditions — Musculoskeletal Diseases; Occupational Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Participatory Organizational Intervention (Experimental): Participatory intervention (workshops) with workers, consultants and leaders. The workshops will find solutions for increased use of assistive devices
  Interventions: Behavioral: Participatory Organizational Intervention
- Control (No Intervention): This group will go through the same baseline and follow-up tests as the intervention group, but will not receive any intervention.

INTERVENTIONS:
Behavioral: Participatory Organizational Intervention
  Arms: Participatory Organizational Intervention

SUMMARY:
Epidemiological studies have shown that patient transfer is a risk factor for back pain, back injuries and long term sickness absence, whereas consistent use of assistive devices during patient transfer is associated with reduced risk of back injury. In consequence, Danish hospitals have made great efforts to increase knowledge, availability and use of assistive devices to reduce work-related physical strain due to patient transfer. Yet, a recent survey among more than 300 nurses and nurses' aides showed that two thirds rarely uses assistive devices during patient transfer. Thus it seems relevant to investigate barriers, opportunities and practical solutions for increasing use of assistive devices among healthcare workers. The purpose of this study is to evaluate a participatory organizational intervention for improved use of assistive devices during patient transfer.

ELIGIBILITY:
At the department level:

Hospital departments with frequent patient handling will be eligible for participation in the cluster-randomized study.

At the individual level (questionnaire replies):

Inclusion Criteria:

* Healthcare workers with daily patient handling (based on questionnaire reply at baseline)

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Use of assistive devices (push-button) | Average use during the entire 1-year follow-up (i.e. continous measurement during 1 year) adjusted for use during 4 weeks prior to the intervention (baseline)
  The healthcare workers are encouraged to push one of the following two buttons every time they leave the room after having performed patient transfer; button 1 "Press this button if you used the necessary assistive devices for your patient transfer" and button 2 "Press this button if you did not use the necessary assistive devices for your patient transfer". The number of Button 1 counts as a percentage of total counts (Button 1+2) will be calculated for set of counters and used as primary outcome.

SECONDARY OUTCOMES:
Use of assistive devices (accelerometer) | change from baseline to 1-year follow-up
  Accelerometers will be placed on the assistive devices. The method is currently being validated in the laboratory and will be finalized before initiation of the 1 year follow-up measurement. Accelerations of a certain time frame will be defined as "use", whereas brief accelerations will be considered as noise
Pain intensity (VAS scale) | change from baseline to 1-year follow-up
  Pain intensity in the low-back is rated subjectively using a 0-10 modified VAS scale, where 0 indicates "no pain at all" and 10 indicate "worst pain imaginable"
Perceived physical exertion (Borg CR10 scale) | change from baseline to 1-year follow-up
  Perceived physical exertion during patient handling. Borg CR10 scale
Back injury | change from baseline to 1-year follow-up
  The specific question reads: "Have you within the last 12 months injured your back during patient transfer? (Think of situation where the pain appeared suddenly and unexpectedly)." The respondent replies "yes" or "no"
Work ability (Index questionnaire) | change from baseline to 1-year follow-up
  The full Work Ability Index questionnaire (Ilmarinen)
Social capital (Questionnaire) | change from baseline to 1-year follow-up
  Questionnaire concerning bonding, bridging, linking A, and linking B social capital (Andersen LL 2015 Scandinavian Journal of Public Health)
Knowledge (Questionnaire) | change from baseline to 1-year follow-up
  Specific questionnaire about knowledge about patients transfer and safety at work
Organizational Readiness to Change (Questionnaire) | change from baseline to 1-year follow-up
  Questionnaire about Organizational Readiness to Change
Use of assistive devices (Questionnaire) | change from baseline to 1-year follow-up
  Questionnaire about frequency of use of the different types of assistive devices

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — National Research Centre for the Working Environment
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Jakobsen MD, Clausen T, Andersen LL. Can a participatory organizational intervention improve social capital and organizational readiness to change? Cluster randomized controlled trial at five Danish hospitals. J Adv Nurs. 2020 Oct;76(10):2685-2695. doi: 10.1111/jan.14441. Epub 2020 Aug 14. PMID 32496600
- [Derived] Jakobsen MD, Aust B, Dyreborg J, Kines P, Illum MB, Andersen LL. Participatory organizational intervention for improved use of assistive devices for patient transfer: study protocol for a single-blinded cluster randomized controlled trial. BMC Musculoskelet Disord. 2016 Dec 20;17(1):501. doi: 10.1186/s12891-016-1339-6. PMID 27998265